CLINICAL TRIAL: NCT00104897
Title: A Phase II Trial to Assess the Activity of 17-allylamino, 17-demethoxygeldanamycin (17-AAG) in Patients With Metastatic (M1, M1b & M1c) Malignant Melanoma
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CRUK-PH2/049; CDR0000415352 (Registry Identifier: PDQ (Physician Data Query)); NCI-6500
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2008-03

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — tanespimycin

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well 17-N-allylamino-17-demethoxygeldanamycin works in treating patients with metastatic malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) in patients with metastatic malignant melanoma.
* Determine the progression-free rate in patients treated with this drug.

Secondary

* Determine the toxicity profile of this drug in these patients.
* Determine the duration of response in patients treated with this drug.
* Determine the survival of patients treated with this drug.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. After 3 courses of treatment, disease response is assessed. Patients with stable or responding disease receive additional courses of treatment.

After completion of study treatment, patients are followed at 28 days and then every 3 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant melanoma

  * Metastatic (M1a, M1b, or M1c) disease
* Measurable disease by clinical exam, x-ray, CT scan, or MRI
* Must have documented disease progression at 2 time points separated by ≥ 6 months

  * Pre-existing visceral lesions or the appearance of new visceral lesions allowed
  * New skin disease amenable to surgery not allowed
* No primary brain tumors or brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin normal
* ALT and AST ≤ 1.5 times upper limit of normal
* No chronic liver disease
* No known hepatitis B or C positivity

Renal

* Creatinine < 130 mmol/L OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No unstable angina pectoris
* No cardiac arrhythmia
* No transient ischemic attack
* No stroke or peripheral vascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 4 weeks before, during, and for 6 months after study participation
* No ongoing or active infection
* No diabetes mellitus with evidence of severe peripheral vascular disease or ulcers
* No history of allergy to eggs
* No known HIV positivity
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other malignancy except adequately treated cone-biopsied carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* More than 4 weeks since prior endocrine therapy
* Concurrent steroids allowed provided they are given at the lowest possible maintenance dose

Radiotherapy

* More than 4 weeks since prior radiotherapy unless administered for palliative care
* Concurrent radiotherapy allowed provided it is administered as a single fraction for bone pain OR as indicated for palliative care

Surgery

* Not specified

Other

* Recovered from all prior therapy

  * Alopecia allowed
* No concurrent therapeutic anticoagulation with warfarin

  * Concurrent prophylactic warfarin for central line maintenance allowed provided INR is checked regularly until stable
  * Concurrent low-molecular weight heparin allowed
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Disease stabilization at 6 months

SECONDARY OUTCOMES:
Toxicity profile as measured by NCI CTCAE version 3
Response duration
Survival
Pharmacodynamic effects as measured by western blot, magnetic resonance spectroscopy, and enzyme-linked immunosorbent assay (ELISA) during course 1
B-RAF and RAS mutation status at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Eisen, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England

REFERENCES:
- [Result] Pacey S, Gore M, Chao D, Banerji U, Larkin J, Sarker S, Owen K, Asad Y, Raynaud F, Walton M, Judson I, Workman P, Eisen T. A Phase II trial of 17-allylamino, 17-demethoxygeldanamycin (17-AAG, tanespimycin) in patients with metastatic melanoma. Invest New Drugs. 2012 Feb;30(1):341-9. doi: 10.1007/s10637-010-9493-4. Epub 2010 Aug 5. PMID 20683637